CLINICAL TRIAL: NCT04780607
Title: Multicenter Results of Mitral Valve Surgery in Patients With Rheumatic Heart Disease
Brief Title: Outcomes of Mitral Valve Surgery in Patients Affected by Rheumatic Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xu Meng, NO.9 department of Cardiac surgery center, Beijing Anzhen Hospital
Other Study IDs: MARS
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-01

CONDITIONS: Outcomes of Mitral Valve Surgery in Patients Affected by Rheumatic Heart Disease
Keywords: rheumtic heart disease; mitral valve surgery
MeSH Terms: interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: mitral valve repair — different repair techniques to construct rheumatic mitral valve lesion

SUMMARY:
rheumatic heart disease remains the majority valvular disease in low and middle income countries, which mostly affected mitral valve, surgical treatment is the most effective strategy to improve the outcomes of middle or late-stage RHD patient, however, whether mitral valve repair surgery is superior to replacement or other evolving interventional device remains controversial, this study aims to investigate the results of repair surgery compared with replacement or other treatment strategy from international multicenters.

ELIGIBILITY:
Inclusion Criteria:

* 1、rheumatic heart disease 2、mitral valve disease 3、combined with other heart valve disease(aortic valve, tricuspid valve, pulmonary valve) 4、patients underwent initial mitral valve surgery or intervention

Exclusion Criteria:

* 1、congenital heart disease degenerative heart valve disease 2、isolated aortic valve or tricuspid valve, pulmonary valve disease( doesn't affect mitral valve ) 3、patients received more than 1 time mitral valve operation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. patients with rheumatic heart disease
  2. mitral valve disease
  3. patients underwent initial mitral valve surgery or intervention
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 2011-2024
  death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: xu meng, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided